CLINICAL TRIAL: NCT06007287
Title: Implementation of World Health Organization Standards for Improving the Quality of Pediatric Hospital Care
Brief Title: WHO Standards for Improving the Quality of Child Hospital Care
Acronym: CHOICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 15/19
Record Dates: First submitted 2023-03-28; First posted 2023-08-23 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-08

CONDITIONS: Pediatric Hospital Care
Keywords: Quality of Care; WHO standards; Children

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Even in high-income countries, quality of pediatric health care has been described as substandard in many settings, resulting in worst health outcomes and increased cost for the health system. Nevertheless, still there is a paucity of studies documenting the quality of care for children in a comprehensive and systematic manner, using international standards, and validated data collection tools. The World Health Organization (WHO) developed three sets standards for improving the quality of maternal newborn and child health care. The aim of this study is to test the use of the WHO Pediatric standards for improving the quality of child hospital care, as summarized by a score of total mean quality score for patients (range 0-100 points).

DETAILED DESCRIPTION:
Achieving the Sustainable Development Goal (SDG) goal 3 targets as elaborated in the WHO Global Strategy for Women's, Children's, and Adolescent's Health (2016-2030) will require ensuring universal access to safe, effective, quality and affordable care for women, children and adolescents. Despite the progress made in the last two decades, an estimated 6.6 million infants, children and young adults still died in 2016 (5.6 million children under five and 1 million children aged 5-14) mostly from preventable causes. To provide universal health coverage with quality, every woman, child and adolescent should receive quality care throughout their life course and during care. This requires institutionalization of safe, effective, quality service delivery.

Studies have shown that most often children do not receive basic elements of care or are often inappropriately managed, and their rights as patients are not respected. Therefore, urgent actions are required to ensure that the care given to all children in health facilities is evidence-based, safe, effective, timely, efficient, equitable and appropriate for their age and stage of development, and that care provided is child and family centred, and that all rights of children are respected. WHO recently launched (May 2018) the "Standards for improving quality of care for children and young adolescents in health facilities", to address the quality of care for children 0-15 years of age in health facilities. These pediatric Standards complement previous standards addressing quality of maternal and newborn care.

The WHO standards are based on a WHO paediatric quality of care framework, which highlights 8 specific domains of care that are critical to providing quality care for children (Fig. 1). These domains are organized into three main categories: provision of care (including: 1. Evidenced based practices; 2. Actionable information system; 3. Functioning referral system), experience of care (including: 4. Effective communication; 5. Respect, protection and fulfilment of child rights; 6. Emotional and psychological support) and availability of child- and adolescent-friendly resources (including 7. Competent, motivated, empathetic human resources and 8. Essential child and adolescent-friendly physical resources). The framework takes into account children's right to health and recognizes that their needs are different from those of adults.

Currently there is very limited field experience in the use of the WHO Standards for improving Quality of Care. More in general, routine use of data to improve case management and organization of care is still not a common practice, even in countries with well-established data collection systems. Despite there are some good examples of how routine data collection systems are used to shape health policies and strategies in the pediatric field in low and middle-income countries, these are quite limited in number, with most of the experience being conducted in a research/project setting.

he aim of this study is to test the use of the WHO Pediatric standards for improving the quality of child hospital care, as summarized by a score of total mean quality score for patients (range 0-100 points).

ELIGIBILITY:
Inclusion Criteria:

* Service Users: parents/ other caretakers of children hospitalised in the Pediatric ward (ordinary hospitalization) and the pediatric emergency unit (brief intensive observation) between 0-15 years in all participating hospital
* Service Providers: all healthcare providers routinely assisting children in the participating units of the hospitals, namely: doctors, doctors in training, nurses

Exclusion Criteria:

Service Users

* Parents/ caretakers with age < 18 years
* Parents/caretakers of a child > 15 years of age (WHO standards cover up to 15 years)
* Parents/ caretakers of deceased child or of a child admitted to intensive care at the time of administration of the questionnaire
* Parents/caretakers with concomitant serious psychiatric disorders
* Parents/caretakers of a child hospitalized at Child Neuropsychiatry or Surgery Department
* Parents/caretakers of a child hospitalized as a Day Hospital
* Parents/caretakers in surgery department/beds of neuro/psychiatric department/beds
* Parents//caretakers with primarily surgery serious psychiatric disorders
* Refusal to participate.

Service Providers

* Personnel not routinely involved in the overall clinical care
* Prolonged absence from work (eg maternity leave) and/or unavailability during the study period
* Personnel working only on surgical conditions or neuro/psychiatric, or other special

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Service users (ie, parents of children hospitalized and their children) and service providers (ie, clinical staff working providing care to children).
Sampling Method: Non-Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Maternal and Newborn Care Index | At hospital discharge (assessed up to day 5)
  Evaluation of total mean quality score for patients (range 0-100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lazzerini, MD, Study Chair — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy